CLINICAL TRIAL: NCT05883566
Title: Comparison of Behavioral , Physiological and Self-reported Pain Responses in Children With Dental Pain
Brief Title: Comparison of Dental Pain Response in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Altamash Institute of Dental Medicine (Other)
Responsible Party: Principal Investigator, Hira Abbasi, Principle investigator, Altamash Institute of Dental Medicine
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: Dental Pain in children
Record Dates: First submitted 2023-05-21; First posted 2023-06-01 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Dental Anxiety

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- behaviour (Experimental)
  Interventions: Behavioral: experimental
- control (No Intervention)

INTERVENTIONS:
Behavioral: experimental — During the procedure, the chairside assistant can capture video recordings of the child's behavior and facial expressions. These videos can be later reviewed by a trained observer who can evaluate the child's pain experience
  Arms: behaviour

SUMMARY:
Study involves the observation of the child's behavior during a dental treatment procedure. This allows for the evaluation of the child's experience of pain and discomfort through their facial expressions, body movements, and vocalizations during the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age range: Children aged between 6-12 years old (or any other specific age range) will be included in the study.
* Dental pain: Participants who have been diagnosed with dental pain by their dentist will be included.
* Consent: Informed consent must be obtained from the child and their parents or guardians before the study.

Exclusion Criteria:

* Participants with existing medical or psychological conditions that could affect the pain response for instance, children with chronic pain conditions or with a history of anxiety or depression.
* Participants who have taken any pain medication within the past 24 hours as this could interfere with the pain response.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Post operative pain | immediately after completion of the treatment within 60 seconds
  Analysis of pain after the treatment pain will be measured by using Visual Analogue Scale(VAS) which is an 10-point scale from 0-10 where 0 represents no pain and 10 represents the worst pain measured

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Hira, Karachi, Sindh
  - Hira Danish, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abbasi H, Saini RS, Binduhayyim RIH, Kuruniyan MS, Mosaddad SA, Heboyan A. Comparison of behavioural, physiological, and self-reported pain responses in Pakistani children with dental pain: a descriptive cross-sectional study. Eur Arch Paediatr Dent. 2025 Dec;26(6):1181-1192. doi: 10.1007/s40368-025-01090-x. Epub 2025 Aug 3. PMID 40753526